CLINICAL TRIAL: NCT01883713
Title: A Prospective Analysis of Methemoglobin as a Biomarker of Tissue Hypoxia During Acute Hemodilutional Anemia in Patients Undergoing Heart Surgery
Brief Title: Study of Methemoglobin as a Biomarker of Tissue Hypoxia During Acute Hemodilution in Heart Surgery Patients
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 12-015
Record Dates: First submitted 2013-03-11; First posted 2013-06-21 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Other Functional Disturbances Following Cardiac Surgery
Keywords: anemia; CPB; methemoglobin; hypoxia
MeSH Terms: conditions — Anemia; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma will be retained for analysis of plasma erythropietin, hepcidin and and nitrate/nitrite levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart surgery during CPB: All patients undergoing heart surgery using cardiopulmonary bypass who have a pre-operative Hb value greater than 90 g/L, no evidence of hypoxemia (SaO2 > 90%) and no history of congenital methemoglobinemia. Exclusion criteria will include severe hypoxemia, acute or chronic renal failure requiring dialysis, emergency surgery or the lack of a PA catheter. Non invasive brain oximetry will be used to assess the brain oxygen tension during surgical procedure.
  Interventions: Device: Brain Oximetry

INTERVENTIONS:
Device: Brain Oximetry — Non invasive brain oximeter will be applied on the patient's forehead to monitor the brain oxygen saturation throughout the surgery.
  Other Names: Nonin equinox oximeter

SUMMARY:
Acute and chronic anemia continue to be associated with increased mortality in a number of clinical settings, including cardiac and non-cardiac surgery. However, "We have no clinical measures that let us know of impending insufficient oxygenation as anemia progresses" (R.B. Weiskopf). The current proposal is based on experimental and clinical data which suggest that plasma methemoglobin (MetHb) may be a sensitive biomarker of tissue hypoxia and "anemic stress" in surgical patients.

Hypothesis: Increased methemoglobin is a biomarker of tissue hypoxia during acute anemia.

Primary Objective: To demonstrate a direct relationship between decreased Hb and increased MetHb in patients undergoing acute hemodilution on cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
Acute and chronic anemia continue to be associated with increased mortality in a number of clinical settings, including cardiac and non-cardiac surgery. 1-6 However, as recently stated by one of the pioneers of anemia research; Dr. R.B. Weiskopf: "We have no clinical measures that let us know of impending insufficient oxygenation as anemia progresses".7 Toward achieving this goal, we have developed experimental models to define the adaptive mechanisms which maintain oxygen homeostasis during acute anemia. Our research has identified that increased nitric oxide (NO) production by nitric oxide syntheses (NOSs) may be an important survival mechanism in acute anemia.3;8;9 Experimental data suggests that nNOS may promote survival by maintaining oxygen (O2) homeostasis during acute anemia.10 Resultant increases in nitric oxide (NO) contributes to adaptive cell signaling mechanisms and also increase oxidation of hemoglobin (Hb) to methemoglobin (MetHb).3 In addition, oxygen extraction results in increased levels of deoxyhemoglobin which has been proposed to act as a nitrite (NO2-) reductase to generate additional bioactive NO, thereby promoting vasodilation in hypoxic vascular beds.11-15 Thus, by more than one mechanism, increased MetHb may be indicative of hemoglobin desaturation, tissue hypoxia and activation of adaptive tissue responses to anemia. These responses may identify the threshold for local tissue hypoxia or "anemic stress". In attempt to determine if such mechanisms are active in humans we performed a retrospective study in patients undergoing cardiopulmonary bypass (CPB) during heart surgery to determine if plasma MetHb increased as Hb decreased during CPB. We observed an inverse relationship between Hb and MetHb that was independent of red blood cell transfusion and exogenous nitrate use

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing heart surgery using cardiopulmonary bypass at St. Michael's Hospital who have a pre-operative Hb value greater than 90 g/L, no evidence of hypoxemia (SaO2 > 90%) and no history of congenital methemoglobinemia.

Exclusion Criteria:

* severe hypoxemia, acute or chronic renal failure requiring dialysis, emergency surgery or the lack of a PA catheter (current standard of care at St. Michael's Hospital is to insert a PA catheter in > 90% of patients).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Arterial methemoglobin levels | 18 months
  To determine if there is an association between increased methemoglobin and tissue hypoxia following heart surgery

SECONDARY OUTCOMES:
Cerebral tissue oxygen saturation | 18 months
Plasma erythropoietin levels | 18 months
Plasma nitrate/nitrite levels | 18 months
Plasma hepcidin levels | 18 months
  Relationship between plasma hepcidin levels and hemoglobin levels

OTHER OUTCOMES:
Adverse outcomes including mortality, myocardial infarction, low output syndrome, stroke and renal dysfunction | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hare, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hare GMT, Han K, Leshchyshyn Y, Mistry N, Kei T, Dai SY, Tsui AKY, Pirani RA, Honavar J, Patel RP, Yagnik S, Welker SL, Tam T, Romaschin A, Connelly PW, Beattie WS, Mazer CD. Potential biomarkers of tissue hypoxia during acute hemodilutional anemia in cardiac surgery: A prospective study to assess tissue hypoxia as a mechanism of organ injury. Can J Anaesth. 2018 Aug;65(8):901-913. doi: 10.1007/s12630-018-1140-0. Epub 2018 Apr 25. PMID 29696581